CLINICAL TRIAL: NCT05193461
Title: The Potential Role of SI00B and Brain Derived Neurotrophic Factor in Predicting Outcome From Using Pulsed Radiofrequency in Treatment of Patients With Lumbar Disc Prolapsed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Wael Fathy Hassan, Assistant Professor of Anaesthesia and pain, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FMBSUREC/06042021/FATHY-2
Record Dates: First submitted 2022-01-02; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Investigation the Role of BDNF and S100B Serum Level as a Predictive of Outcome of Pulsed Radiofrequency in Treatment Lumbar Disc Prolapse Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with radicular pain recieved pulsed mood radiofrequency (Experimental): Investigation effect of neuroplasticity of patient on outcome of pulsed mood radiofrequency
  Interventions: Procedure: Pulsed mood radiofrequency on dorsal root ganglion

INTERVENTIONS:
Procedure: Pulsed mood radiofrequency on dorsal root ganglion — 3) Pulsed radio frequency (PRF): PRF of the dorsal root ganglion (DRG) will be performed to all participants in this study. The procedures will be performed in the operating room under fluoroscopic guidance following radiation safety standards. The dorsal root ganglion of lumbosacral roots will be targeted. The patients will be positioned prone .Lidocaine 1% will be infiltrated at the skin entry site. A 10 cm, 22-gauge radiofrequency needle with a 5 mm curved active tip will be used. A radiculogram will be done to confirm appropriate placement and DRG will be stimulated for confirmation of the appropriate nerve root involved. Proximity of the needle to the DRG will be determined by appropriate sensory stimulation with 50 Hz (0.4-0.6 V), and motor stimulation at 2 Hz will be used to determine a threshold 1.5-2.0 times greater than the sensory threshold to avoid placement near the anterior nerve root. A pulsed lesion will be generated by applying 45 V to the DRG for 6 minutes at 42°C.

SUMMARY:
Chronic lumbar radicular (CLR) pain is a term used to describe neuropathic pain symptoms in the distribution of a particular lumbar nerve root due to disc protrusion, spinal stenosis, facet hypertrophy, or fibrosis after previous surgery. The pathophysiology of CLR pain involves mechanical, inflammatory, and immunologic factors that affect the function of the dorsal root ganglion (DRG).1Treatment methods include oral pain medications, physical therapy, epidural steroid injection (ESI) and surgery. 2,3.

Pulsed radiofrequency (PRF) was developed as a modification of the well-known radiofrequency ablation treatment. In conventional radiofrequency ablation, a high frequency alternating current is used to produce coagulative necrosis of the target nerve tissue without any selectivity for nociceptive fibers. However, in PRF, a current in short (20 msec) high voltage bursts is followed by silent phases (480 msec) which allow for heat dissemination, keeping the target tissue controlled below 42°C. 4,5 The mechanisms via which PRF causes analgesia are still not clearly understood, but laboratory experiments have highlighted some possible ways in which it might act, including its effects on neuropathic pain. Clinical use of PRF has been expanding, despite there being limited evidence of clinical efficacy in the form of randomized controlled trials (RCTs). 6 There have been few RCTs using PRF-DRG for radicular pain. Van Zundert et al performed an RCT in subjects with cervical radicular pain.7 Simopoulos et al did a pilot study on lumbar radicular pain, but the methodology included application of conventional radiofrequency over PRF in the study group and was not an efficacy trial. As such, the efficacy of PRF-DRG in CLR has never been determined. 8

Neuroplasticity or neuronal plasticity refers to the ability of the nervous system to do neuronal remodeling, formation of novel synapses and birth of new neurons. Neuronal plasticity is intimately linked to cellular responsiveness and may therefore be considered an index of the neuronal capability to restore its function. Failure of such mechanisms might enhance the susceptibility to neuronal injury.9 Neurotrophic factors (NTFs), and in particular the neurotrophin family, play an important role. In fact, besides their classical role in supporting neuronal survival, NTFs finely modulate all the crucial steps of network construction, from neuronal migration to experience-dependent refinement of local connections. It is now well established that NTFs are important mediators of neuronal plasticity also in adulthood where they modulate axonal and dendritic growth and remodeling, membrane receptor trafficking, neurotransmitter release, synapse formation and function.10 The neurotrophin brain-derived neurotrophic factor (BDNF) has emerged as crucial mediator of neuronal plasticity, suggesting that it might indeed bridge experience with enduring change in neuronal function.11BDNF acts on certain neurons of the central nervous system and the peripheral nervous system, helping to support survival of existing neurons, and encouraging growth and differentiation of new neurons and synapses.12,13 S100B belongs to the family ofcalcium binding proteins, is expressed mainly by astrocytesand is found both intra- and extracellularly in brain tissue. It was also reported that mature myelinating and non-myelinating Schwann cells of peripheral nerves strongly display S100 protein immunoreactivity (Stefansson et al., 1982; Sugimura et al., 1989; Vega et al., 1996).14 S100B can spill from injured cells and enter the extracellular space or bloodstream. Serum levels of S100B increase in patients with neuronal damage. Over the last decade, S100B has emerged as a candidate peripheral biomarker of neuronal injury. Elevated S100B levels accurately reflect the presence ofneurodegenerayion. Its potential clinical use in the therapeutic decisions is substantiated by a vast body of literature. Thus, the major advantage of using S100B is that its elevatio in serum provides a sensitive measure for determining neuronal injury at the molecular level before gross changes level.15

DETAILED DESCRIPTION:
METHODS:

All patientswill be subjected to the following:

1) Clinical assessment:

1. Detailed history taking regarding: duration of pain, the presence of discogenic pain, radicular pain, responseto medical treatment, or previous interventional pain management
2. Neurological examination: motor and sensory examination
3. Assessment of the severity of the neurological symptoms before, 2 week, 1, 3 and 6 months after the interventional procedure by a physician who will be blinded to the patient's condition and the type of intervention.

   Modified Oswestry Back Disability Score (MODI): It consisted of low back pain disability index questionnaire about pain intensity, personal care, lifting, standing, walking, sitting, sleeping, social life, travelling and employment/homemaking. Thus, total 10 points; each had score range of 0-5. Hence, total score had range of 0-50. A high MODI score indicates a more severe functional disability related to the pain.

   Numeric Rating Scale (NRS-11): It is a scale for assessment of intensity of pain. It ranged from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain.
4. Assessment of patient's satisfaction about the intervention,2 week, 1, 3, and 6months after the interventional procedure by a physician who will be blinded to the patient's condition and the type of intervention.

The Short Assessment of Patient Satisfaction (SAPS): It consists of seven items assessing the core domains of patient satisfaction which include treatment satisfaction, explanation of treatment results, clinician care, participation in medical decision making, respect by the clinician, time with the clinician, and satisfaction with hospital/clinic care. Responses scales are 5-point scales. SAPS scores can be interpreted as follows: 0 to 10 = very dissatisfied, 11 to 18 = dissatisfied, 19 to 26 = satisfied, 27 to 28 = very satisfied.

2) Radiological assessment:

Magnetic Resonance imaging (MRI):

Magnetic Resonance imaging of the lumbosacral spine will be performed for all patients included in the study.

The following protocols will be used:

1. T1- weighted images (axial, sagittal).
2. T2- weighted images (axial, coronal).
3. Fluid attenuated inversion recovery (FLAIR) sequence. 3) Pulsed radio frequency (PRF): PRF of the dorsal root ganglion (DRG) will be performed to all participants in this study. The procedures will beperformed in the operating room under fluoroscopic guidance following radiation safety standards. The dorsal root ganglion of lumbosacral roots will be targeted. The patients will be positioned prone .Lidocaine 1% will be infiltrated at the skin entry site. A 10 cm, 22-gauge radiofrequency needle with a 5 mm curved active tip will be used. A radiculogram will be done to confirm appropriate placement and DRG will be stimulated for confirmation of the appropriate nerve root involved. Proximity of the needle to the DRG will be determined by appropriate sensory stimulation with 50 Hz (0.4-0.6 V), and motor stimulation at 2 Hz will be used to determine a threshold 1.5-2.0 times greater than the sensory threshold to avoid placement near the anterior nerve root. A pulsed lesion will be generated by applying 45 V to the DRG for 6 minutes at 42°C.

4) Laboratory assessment

A. Assessment of Brain Derived Neurotrophic Factor (BDNF) serum level:

Venous blood samples will be taken from all included patients before the interventional procedure and kept 30 minutes for clotting then centrifuged at 2,000-3,000 rpm for 20 minutes. Then, serum will be separated and kept under -80 c. The BDNF levels will be assessed using commercial sandwich-ELISA kits. The Microelisastripplatewill be pre-coated with an antibody specific to BDNF. Samples will be added to the appropriate Microelisastripplate wells and comoned to specific antibody. Then a Horseradish Peroxidase (HRP) conjugated antibody specific for BDNF will be added to each 'Microelisastripplate well and incubated. Free components will be washed away. The TMB substrate solution will be added to each well. Only those wells that contain BDNF and HRP conjugated BDNF antibody will appear blue and then turn to yellow after the addition of the stop solution. The optical density (OD) will be measured spectrophotometrically at a wavelength of 450 nm.

B. Assessment of S100B serum level:

All participants will undergo quantitative assessment of serum S100B before the interventional procedure by applying a sandwich enzyme- linked immunoabsorbent assay technique (ELISA). Assays will be performed at the clinical and chemical pathology department, Beni-suef university hospital on an automated ELISA platform. Five mL of whole blood will be drawn from all included patients and put into a sterile plain tube. The blood samples will be centrifuged for twenty minutes at a speed 2000-3000 r.p.m. The supernatant serum will be collected and stored at -20 C till the time of analysis. Standard of S100B will be supplied as 120 microlitre containing 4000ng/L of S100B diluted by standard diluents to generate dilution range from 0 to 2000ng/L. Fifty mL of standard will be added to wells, they will be incubated for one hour at room temperature. The wells will be washed three times with washing solution (phosphate buffered saline, PH is from 7.0 to 7.2). 100 mL of conjugate will be added per each well. Each well will be washed again by washing solution five times. Fifty mL of substrate A (S100B horseradish peroxidase (HRP) conjugate) will be added to each well followed by addition of Fifty mL of substrate B (substrate for HRP enzyme containing small amount of 3,3,5,5 tetramethylbenzidine) then the wells will be covered and left at room temperature for ten minutes. Finally, fifty mL of stop solution (sulphuric acid) will be added to each well. Optical density will be read at 450 nm. The standard curve will be constructed using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having symptomatic lumbar disc prolapse based on the following:

  1. Clinical evidence of disc pulge in the form of disc related radicular pain of >3 months duration with failed conservative treatment (i.e. physical therapy and multiple medications) and unwillingness to pursue surgical option.
  2. Radiological demonstration of posterolateral lumbar disc pulge by MRI or CT lumbosacral
  3. Age range is between 30-80 years

Exclusion Criteria:

* The following patients will be excluded from the study:

  1. Patients with spinal deformities
  2. Patients with a previous history of spinal trauma
  3. Patients with radiological evidence of any inflammatory or neoplastic lesion affecting the spinal cord or vertebral column
  4. Patients with severe lumbar disc herniation causing lower limb weakness or sphincteric troubles
  5. Patients with contraindications to interventions (coagulopathy or sepsis)
  6. Patients with contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body).
  7. Pregnant

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The functional outcome from using pulsed radiofrequency in treatment of patients with lumbar disc prolapse | 6 months
  Pre intervention serum BDNF

SECONDARY OUTCOMES:
The functional outcome from using pulsed radiofrequency in treatment of patients with lumbar disc prolapse | 6 months
  Pre intervention serum S100B

CONTACTS AND LOCATIONS:
Locations (1):
- Wael Fathy Hassan, Banī Suwayf, Egypt